CLINICAL TRIAL: NCT03410745
Title: The Effect of Exercise on the Collagen Synthesis and Cytokine Response in Human Cartilage Tissue With Osteoarthritis
Brief Title: Cartilage Adaptation and Response to Interleukins and Exercise
Acronym: CARTILEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Adam El Mongy Jørgensen, MD, Principal Investigator, Medical Doctor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BBH-139
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Osteo Arthritis Knee
Keywords: exercise; cytokines; collagen
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental)
  Interventions: Behavioral: Exercise.
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Exercise. — Moderate to heavy intensity resistance exercise consisting of leg press.
  Arms: Exercise group

SUMMARY:
This study will examine the effect of exercise on the turnover of collagen in articular cartilage and the content of cytokines in the synovial fluid from human adults with osteoarthritis.

DETAILED DESCRIPTION:
By using stabile isotope labelling, this study will track the formation and destination of newly formed cartilage collagen in adult humans scheduled for knee replacement surgery due to osteoarthritis. The collagen formation as well as the effect on the cytokine content of the synovial fluid will be examined both at rest and in response to 4 weeks of exercise/training. Overall the project aims to improve the basic understanding of cartilage development and function in relation to osteoarthritis prevention.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of the knee scheduled for knee replacement surgery
* Must be able to perform physical exercise
* Age 40-90 years old
* BMI 18.5-40 kg/m^2
* None smoker for the last 6 weeks

Exclusion Criteria:

* Regular intake of:
* non steroid anti-inflammatory drugs (NSAID)
* corticoid-steroids
* disease modifying anti-rheumatic drugs (DMARD)
* cytostatic incl. chemotherapy
* immune suppressive medicine
* Inflammatory diseases or cancer
* Recent trauma to the knee (< 3 months)
* Previous knee surgery
* Regular strenuous exercise ( > 1 pr. month)
* Previous exposure to tracers (e.g. from another study)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Collagen synthesis in articular cartilage | End of study at 4 weeks
  By using incorporation of stabile isotope tracers measured by gas chromatography, the concentration of newly formed collagen will be measured.

SECONDARY OUTCOMES:
Cytokine and enzymes concentration in synovial fluid | End of study at 4 weeks
  By using Enzyme-Linked Immunosorbent Assay (ELISA) the concentration of cytokines in synovial fluid will be measured.
Cytokine and enzymes concentration in blood | At the beginning and at the end of the study at 4 weeks
  By using Enzyme-Linked Immunosorbent Assay (ELISA) the concentration of cytokines in the blood will be measured.
Gene expression | End of study at 4 weeks
  By using real time reverse transcriptase polymerase chain reaction (RT-PCR) the concentration of messenger ribonucleic acid (mRNA) in cartilage tissue will be measured.
Strength | At the beginning and at the end of the study at 4 weeks
  By calculating the total volume of weight lifted (kg) the strength will be measured.
Body mass index (BMI) | At the beginning of the study.
  BMI measured as the total body weight divided by the height squared (kg/m^2)
Age | At the beginning of the study.
  The age measured in years

CONTACTS AND LOCATIONS:
Overall Officials: Adam EM Jørgensen, MD, Principal Investigator — Institute of Sports Medicine, Copenhagen
Locations (1):
- Institute of Sports Medicine Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Jorgensen AEM, Schjerling P, DellaValle B, Rungby J, Kjaer M. Acute loading has minor influence on human articular cartilage gene expression and glycosaminoglycan composition in late-stage knee osteoarthritis: a randomised controlled trial. Osteoarthritis Cartilage. 2023 Jul;31(7):884-893. doi: 10.1016/j.joca.2023.01.317. Epub 2023 Jan 30. PMID 36720425